CLINICAL TRIAL: NCT06928909
Title: Evaluating the Feasibility of an Intensity-Adapted Pediatric Acute Myeloid Leukemia Treatment Guideline in Malawi
Brief Title: Leukemia Adapted Protocol
Acronym: LEAP
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: American Society of Hematology (Other)
Responsible Party: Principal Investigator, Casey McAtee, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-53055
Record Dates: First submitted 2025-03-19; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Pediatric Acute Myeloid Treatment; Acute myeloid leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients with de novo AML: All patients with de novo AML presenting to Kamuzu Central Hospital in Lilongwe, Malawi will be offered enrollment into the study.
  Interventions: Other: Intensity-adapted pediatric acute myeloid treatment guidelines

INTERVENTIONS:
Other: Intensity-adapted pediatric acute myeloid treatment guidelines — This is an observational study evaluating the current standard of care AML therapy in Malawi. The therapy guideline used is an adaptation of the International Society of Paediatric Oncology (SIOP) guidelines for pediatric AML in resource-constrained centers published by the International Society of Paediatric Oncology (SIOP). It is currently the standard of care in Malawi for all patients with AML. Receipt of this therapy guideline is independent of participation in research.

SUMMARY:
In resource-constrained settings such as Malawi, survival rates for pediatric acute myeloid leukemia (AML) are dismally low compared to high-resource environments. This disparity highlights the urgent need for feasible treatment protocols tailored to the realities of these regions where most children with cancer are treated. In 2023, after reviewing favorable clinical trials results in other resource-limited settings, the Kamuzu Central Hospital (KCH) pediatric cancer unit adopted an evidence-based intensity-adapted clinical practice guideline (CPG) developed by the International Society of Paediatric Oncology (SIOP) as its standard of care for the treatment of pediatric AML, aiming to balance curative intent with manageable toxicity. The current study is a prospective evaluation of outcomes of standard of care in Malawi using the SIOP CPG in a real-world setting.

The LEAP study aims to assess the implementation of the SIOP AML guidelines at KCH in an effort to continually improve outcomes in Malawi. The study is an observational-implementation design with a composite effectiveness-implementation outcome called Implementation Success. Implementation Success combines feasibility, the ability of patients to complete all aspects of the CPG, with effectiveness, the ability to maintain historical rates of complete remission of 40% at the treatment center.

This prospective cohort study will enroll children under 18 years diagnosed with de novo AML at KCH. Implementation Success will be the primary endpoint, with secondary endpoints including CPG fidelity, long-term survival, adverse events, and hematologic recovery times. Patient-reported outcomes will also be collected to assess the impact of treatment on quality of life.

This will be the first prospective study of pediatric AML in sub-Saharan Africa, providing critical data on the management of AML in low-resource settings. By assessing the implementation of a context-adapted CPG, the study will contribute to the global effort to improve pediatric AML outcomes in resource-constrained environments. The findings will serve to guide practitioners in Malawi and similar settings, and the data generated will be invaluable for future clinical decisions and CPG development.

DETAILED DESCRIPTION:
Participants:

* All patients with have de novo AML presenting to Kamuzu Central Hospital (KCH) in Lilongwe, Malawi will be offered enrollment into the study.
* Patients must be <18 years of age at time of study enrollment.
* Patients must begin treatment according to the 2023 KCH AML therapy CPG.
* All patients at the treating center receiving curative-intent therapy for AML are treated on the 2023 KCH AML standard of care CPG based on the SIOP AML guidelines, independent of participation in research.
* Patients should ideally be consented for data collection within one week of confirmatory diagnosis to ensure highest quality of prospective data collection.

The therapy guideline used at KCH is based upon the published international guidelines for treating pediatric AML in resource-constrained centers published by the International Society of Paediatric Oncology (SIOP). It is currently the standard of care at KCH.

Data Collection Schedule:

All study measurements in this study are routinely captured as part of clinical care. No additional clinical studies will be obtained from patients as a consequence of enrollment onto the LEAP study.

1. On-treatment schedule Patients are routinely admitted inpatient to the pediatric cancer unit at the start of each chemotherapy cycle. Patients remain inpatient according to standard practices of the unit until they no longer require routine blood product transfusions and their absolute neutrophil count is rising. Patients are discharged home for ~1 week prior to returning to start the subsequent cycle, but generally no later than 2 weeks from discharge.

   Required Data Items are all routinely obtained as part of standard of care:
   * Bone marrow aspirate with morphology +/- trephine biopsy
   * Bone marrow flow cytometry OR immunohistochemistry
   * Lumbar puncture with cerebrospinal fluid cell count & morphological evaluation
   * Leukemia cytogenetics
   * Lanksy score
   * Weight, height, MUAC
   * History & physical
   * Complete blood count
   * Serum electrolytes
   * Confirmation of HIV serostatus (standard of care for all pediatric patients in Malawi)
   * Chest X-ray
   * Echocardiogram
   * Adverse event monitoring
   * PROMIS-25 parent & patient questionnaire (additional research-only evaluation)
   * REDCap data upload
2. Post-treatment schedule Patients will be followed up by telephone monthly for the first six months off therapy. In-person visits routinely occur at 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months following completion of therapy. They are followed annually thereafter.

Required Data Items:

* History and confirmation of vital status
* Physical exam
* Complete/full blood count
* PROMIS-25 questionnaire
* REDCap data upload

Statistical analysis:

Sample size determination of this study is based on accrual capacity of the study site, not from statistical power. Based on diagnoses over the previous three years at Kamuzu Central Hospital in Malawi, the investigators expect at least 10 de novo cases/year of AML.

Primary Endpoint

CPG Implementation Success will be a composite endpoint comprised of:

1. Feasibility: proportion of patients completing the CPG
2. Effectiveness: proportion of patients in complete remission (CR) by the end of Induction

Implementation will be deemed successful if 1) ≥50% of patients are able to complete the CPG; AND 2) The historical benchmark of end-of-induction complete remission (CR) of 40% is maintained.

Rates of CR (effectiveness outcome) and CPG completion (implementation outcome) will be monitored continuously by the study statistician team using an adaptation of the method of Ivanova and colleagues. This method provides a Pocock-type boundary so that the probability of crossing the boundary is at most 5% when the true rate of the event crosses the acceptable threshold. For the effectiveness threshold of CR, we will use the established historical rate of CR of 40% achieved on the old standard of care for AML in Malawi. The probability of boundary crossing rises to 24%, 68%, and 98% if the CR rate drops to 30%, 20%, and 10%, respectively, with corresponding accruals of N=28, 22, and 14. Similarly, for rate of CPG completion, we will use a threshold of 50%. The probability of boundary crossing rises to 22%, 59%, and 92% if the rate of completion rate drops to 40%, 30%, and 20%, respectively, with corresponding expected accruals of N=27, 22, and 15.

Criteria for completing the CPG are:

1. Completing all required chemotherapy cycles (Induction 1, Induction 2, Consolidation 1, Consolidation 2) and achieving transfusion independence following Consolidation 2 outside of the setting of relapse or bone marrow failure (in which case therapy will be considered complete for the purposes of the study outcome). Note that pre-phase is not required for completion.
2. Completion of Inductions 1 and 2 but not in CR at the end of Induction.
3. Completion of Inductions 1 and 2 having achieved CR by the end of Induction 2 but having had relapse prior to completing Consolidation 2.
4. All patients with early mortality (≤42 days), treatment-related mortality, or treatment abandonment of curative-intent therapy will be considered incomplete.
5. Patients removed from curative-intent therapy due to toxicity will be considered incomplete.

Complete Remission is defined as <5% myeloblasts on bone marrow evaluation.

Secondary Endpoints

* Event-free, relapse-free, and overall survival at 12 & 24 months from diagnosis
* Proportion of patients with CTCAE ≥3 adverse events
* Patient-reported outcomes at diagnosis, end of induction, end of therapy, and 6 months post-therapy.
* Cytogenetic characteristics of myeloblasts
* Proportion of discrete treatment and supportive care CPG elements received/completed as prescribed

ELIGIBILITY:
Inclusion Criteria:

1. Age Patients must be <18 years of age at time of study enrollment.
2. Diagnosis

   Patients must be diagnosed with de novo AML according to 2022 WHO 5th Edition classification with or without extramedullary disease. Patients must have one of the following:
   * Bone marrow myeloblasts ≥20%. In cases of dry taps due to fibrosis, myeloblast percentage can be estimated from a bone marrow biopsy core specimen. Due to unavailable molecular/cytogenetic diagnostics in Malawi, patients with <20% bone marrow myeloblasts can be included in the study at the discretion of the treating oncologist with rationale documented.
   * In cases where a bone marrow evaluation is not safe/feasible, a peripheral blood sample may be used with a documented absolute myeloblast percentage of ≥1000/μL calculated based on a total white blood cell count and percentage circulating blasts.
3. Therapy Patients must begin treatment according to the 2023 KCH AML therapy CPG.

Exclusion Criteria:

1. Patients with any of the following conditions or criteria will be excluded from the study:

   * Juvenile myelomonocytic leukemia
   * Transient myeloproliferative disorder
   * Acute promyelocytic leukemia
   * Mixed phenotype acute leukemia
   * Trisomy 21
   * Current pregnancy
   * Previous or concurrent malignancy
   * Isolated myeloid sarcoma
2. Patients previously treated with antineoplastic therapy with the following exceptions:

   * Hydroxyurea
   * Corticosteroids
   * Intrathecal chemotherapy at diagnosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients with de novo AML presenting to Kamuzu Central Hospital in Lilongwe, Malawi.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the implementation success of an intensity adapted clinical practice guideline (CPG) based upon recommendations by the International Society of Paediatric Oncology (SIOP) for childhood AML in resource limited settings. | From initiation of chemotherapy to assessment of completion of the CPG and attainment of end-of-induction bone marrow evaluation (if CPG completed to that point), assessed up to 12 months from the start of chemotherapy.
  CPG Implementation Success will be a composite endpoint comprised of:
  1. Feasibility: proportion of patients completing the CPG. (see Study Design for further details outlining CPG completion criteria)
  2. Effectiveness: proportion of patients in complete remission (CR) by the end of Induction 2 chemotherapy.

SECONDARY OUTCOMES:
Estimate the proportion of patients with negative minimal residual disease (MRD) following Induction | By end of second induction, assessed up to 6 months from initiating chemotherapy.
  MRD will be evaluated by bone marrow examination with multiparameter flow cytometry. MRD positivity will be defined as ≥0.1% residual pathological myeloblasts.
Estimate the proportion of patients with early mortality | Assessed up to 42 days from start of chemotherapy
  Early mortality is defined as death occurring ≤42 days from the beginning of treatment.
Estimate the proportion of patients with treatment-related mortality on the CPG | Assessed from Day 43 following initiation of chemotherapy through to completion of the CPG, assessed up to 12 months.
  TRM will be defined as death occurring >42 days from the beginning of treatment due to any cause in the absence of progressive cancer.
Estimate the proportion of patients with serious adverse events | From initiation of chemotherapy through to completion of the CPG, assessed up to 12 months.
  All adverse events among patients treated on the CPG will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5. All the Grade ≥3 adverse events will be recorded
Estimate the time to hematologic recovery following cycles of chemotherapy | From the final dose of curative-intent chemotherapy to blood product independence, assessed up to 6 months.
  Time to transfusion independence of blood products following completion of therapy.
Estimate the proportion of patients with treatment abandonment. | From initiation of chemotherapy to completion of the CPG, assessed up to 12 months.
  After starting Day 1 of therapy, any unplanned hiatus of curative-intent therapy lasting ≥4 weeks lasting ≥4 weeks.
Estimate survival of patients treated with the CPG. | Assessed 24 months from start of therapy
  Overall, event-free, and relapse-free survival 12 & 24 months from diagnosis.
Describe myeloblast cytogenetics | Time of diagnosis (samples are batched and assessed up to 6 months following diagnostic bone marrow evaluation)
  Myeloblast cytogenetics is defined as reported by NanoString bone marrow analysis at diagnosis.
Describe Patient Reported Outcomes at relevant timepoints. | Assessed within 30 days of diagnostic bone marrow evaluation (diagnosis timepoints) and within 30 days of the end of second induction (mid-therapy time-point, assessed up to 6 months from diagnosis).
  Patient-Reported Outcomes Measurement Information System (PROMIS-25) questionnaires will be given to parents and children enrolled on study at the time of diagnosis (within 30 days) and at the end of second Induction (within 30 days). Questionnaires will be administered by study personnel while patients are inpatient. As many families at the treatment center are illiterate, all questionnaires will be read and filled in by study personnel based on answers by the parents/children.
Determine the fidelity to treatment and supportive care practice guidelines associated with AML therapy in Malawi | From initiation of chemotherapy through to completion of the CPG, assessed up to 12 months.
  Proportion of discrete treatment and supportive care guideline elements received/completed as prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Casey McAtee, M.D., M.P.H., Principal Investigator — Baylor College of Medicine
Locations (1):
- Kamuzu Central Hospital, Lilongwe, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No
Malawian data privacy laws prohibit open sharing of individual patient data. Aggregated data supporting study outcomes will be published as a scientific manuscript. Requests for IPD will be considered on a case-by-case basis by study investigators, following all applicable Malawian data privacy laws.

REFERENCES:
- [Background] Banavali, S. D. et al. PRET: an effective oral protocol for out-patient therapy in patients with acute myeloid leukemia. International Society of Paediatric Oncology Meeting Abstracts (2004).
- [Background] Malani D, Murumagi A, Yadav B, Kontro M, Eldfors S, Kumar A, Karjalainen R, Majumder MM, Ojamies P, Pemovska T, Wennerberg K, Heckman C, Porkka K, Wolf M, Aittokallio T, Kallioniemi O. Enhanced sensitivity to glucocorticoids in cytarabine-resistant AML. Leukemia. 2017 May;31(5):1187-1195. doi: 10.1038/leu.2016.314. Epub 2016 Nov 11. PMID 27833094
- [Background] Tsukimoto I, Tawa A, Horibe K, Tabuchi K, Kigasawa H, Tsuchida M, Yabe H, Nakayama H, Kudo K, Kobayashi R, Hamamoto K, Imaizumi M, Morimoto A, Tsuchiya S, Hanada R. Risk-stratified therapy and the intensive use of cytarabine improves the outcome in childhood acute myeloid leukemia: the AML99 trial from the Japanese Childhood AML Cooperative Study Group. J Clin Oncol. 2009 Aug 20;27(24):4007-13. doi: 10.1200/JCO.2008.18.7948. Epub 2009 Jul 20. PMID 19620491
- [Background] Organization, W. H. World Cancer Day 2023: Message of the WHO Regional Director for Africa, Dr. Matshidiso Moeti. https://www.afro.who.int/regional-director/speechesmessages/ world-cancer-day-2023 (2023).
- [Background] Van Weelderen RE, Klein K, Natawidjaja MD, De Vries R, Kaspers GJ. Outcome of pediatric acute myeloid leukemia (AML) in low- and middle-income countries: a systematic review of the literature. Expert Rev Anticancer Ther. 2021 Jul;21(7):765-780. doi: 10.1080/14737140.2021.1895756. Epub 2021 Mar 29. PMID 33779466
- [Background] Roberts N, James S, Delaney M, Fitzmaurice C. The global need and availability of blood products: a modelling study. Lancet Haematol. 2019 Dec;6(12):e606-e615. doi: 10.1016/S2352-3026(19)30200-5. Epub 2019 Oct 17. PMID 31631023
- [Background] Cooper TM, Absalon MJ, Alonzo TA, Gerbing RB, Leger KJ, Hirsch BA, Pollard J, Razzouk BI, Aplenc R, Kolb EA. Phase I/II Study of CPX-351 Followed by Fludarabine, Cytarabine, and Granulocyte-Colony Stimulating Factor for Children With Relapsed Acute Myeloid Leukemia: A Report From the Children's Oncology Group. J Clin Oncol. 2020 Jul 1;38(19):2170-2177. doi: 10.1200/JCO.19.03306. Epub 2020 May 13. PMID 32401633
- [Background] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Background] Einstein MH, Ndlovu N, Lee J, Stier EA, Kotzen J, Garg M, Whitney K, Lensing SY, Tunmer M, Kadzatsa W, Palefsky J, Krown SE. Cisplatin and radiation therapy in HIV-positive women with locally advanced cervical cancer in sub-Saharan Africa: A phase II study of the AIDS malignancy consortium. Gynecol Oncol. 2019 Apr;153(1):20-25. doi: 10.1016/j.ygyno.2019.01.023. Epub 2019 Feb 15. PMID 30773222
- [Background] Health, N. I. of. Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0. httpsctep.cancer.govprotocolDevelopmentelectronicapplicationsctc.htm (2017).
- [Background] Alexander S, Pole JD, Gibson P, Lee M, Hesser T, Chi SN, Dvorak CC, Fisher B, Hasle H, Kanerva J, Moricke A, Phillips B, Raetz E, Rodriguez-Galindo C, Samarasinghe S, Schmiegelow K, Tissing W, Lehrnbecher T, Sung L; International Pediatric Oncology Mortality Classification Group. Classification of treatment-related mortality in children with cancer: a systematic assessment. Lancet Oncol. 2015 Dec;16(16):e604-10. doi: 10.1016/S1470-2045(15)00197-7. PMID 26678213
- [Background] Creutzig U, van den Heuvel-Eibrink MM, Gibson B, Dworzak MN, Adachi S, de Bont E, Harbott J, Hasle H, Johnston D, Kinoshita A, Lehrnbecher T, Leverger G, Mejstrikova E, Meshinchi S, Pession A, Raimondi SC, Sung L, Stary J, Zwaan CM, Kaspers GJ, Reinhardt D; AML Committee of the International BFM Study Group. Diagnosis and management of acute myeloid leukemia in children and adolescents: recommendations from an international expert panel. Blood. 2012 Oct 18;120(16):3187-205. doi: 10.1182/blood-2012-03-362608. Epub 2012 Aug 9. PMID 22879540
- [Background] Khoury JD, Solary E, Abla O, Akkari Y, Alaggio R, Apperley JF, Bejar R, Berti E, Busque L, Chan JKC, Chen W, Chen X, Chng WJ, Choi JK, Colmenero I, Coupland SE, Cross NCP, De Jong D, Elghetany MT, Takahashi E, Emile JF, Ferry J, Fogelstrand L, Fontenay M, Germing U, Gujral S, Haferlach T, Harrison C, Hodge JC, Hu S, Jansen JH, Kanagal-Shamanna R, Kantarjian HM, Kratz CP, Li XQ, Lim MS, Loeb K, Loghavi S, Marcogliese A, Meshinchi S, Michaels P, Naresh KN, Natkunam Y, Nejati R, Ott G, Padron E, Patel KP, Patkar N, Picarsic J, Platzbecker U, Roberts I, Schuh A, Sewell W, Siebert R, Tembhare P, Tyner J, Verstovsek S, Wang W, Wood B, Xiao W, Yeung C, Hochhaus A. The 5th edition of the World Health Organization Classification of Haematolymphoid Tumours: Myeloid and Histiocytic/Dendritic Neoplasms. Leukemia. 2022 Jul;36(7):1703-1719. doi: 10.1038/s41375-022-01613-1. Epub 2022 Jun 22. PMID 35732831
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] bank, W. World Bank Country Data - Malawi. https://data.worldbank.org/country/MW (2021).
- [Background] GBD 2017 Childhood Cancer Collaborators. The global burden of childhood and adolescent cancer in 2017: an analysis of the Global Burden of Disease Study 2017. Lancet Oncol. 2019 Sep;20(9):1211-1225. doi: 10.1016/S1470-2045(19)30339-0. Epub 2019 Jul 29. PMID 31371206
- [Background] Painschab MS, Westmoreland KD, Kasonkanji E, Zuze T, Kaimila B, Waswa P, El-Mallawany NK, Tomoka T, Mulenga M, Montgomery ND, Fedoriw Y, Gopal S. Prospective study of Burkitt lymphoma treatment in adolescents and adults in Malawi. Blood Adv. 2019 Feb 26;3(4):612-620. doi: 10.1182/bloodadvances.2018029199. PMID 30796065
- [Background] Chakumatha E, Weijers J, Banda K, Bailey S, Molyneux E, Chagaluka G, Israels T. Outcome at the end of treatment of patients with common and curable childhood cancer types in Blantyre, Malawi. Pediatr Blood Cancer. 2020 Jul;67(7):e28322. doi: 10.1002/pbc.28322. Epub 2020 May 11. PMID 32391955
- [Background] Kasonkanji E, Kimani S, Skiver B, Ellis G, Seguin R, Kaimila B, Tomoka T, Mulenga M, Montgomery N, Fedoriw Y, Gopal S, Westmorland KD, Painschab MS. Clinical Characteristics and Outcomes of Acute Lymphoblastic Leukemia in Adolescents and Young Adults in Malawi. JCO Glob Oncol. 2022 Jun;8:e2100388. doi: 10.1200/GO.21.00388. PMID 35772043
- [Background] Rubagumya F, Xu MJ, May L, Driscoll C, Uwizeye FR, Shyirambere C, Larrabee K, Fehr AE, Gilbert UD, Muhayimana C, Hategekimana V, Elmore S, Mpunga T, Moore M, Shulman LN, Lehmann L. Outcomes of Low-Intensity Treatment of Acute Lymphoblastic Leukemia at Butaro Cancer Center of Excellence in Rwanda. J Glob Oncol. 2018 Sep;4:1-11. doi: 10.1200/JGO.2017.009290. Epub 2017 Oct 30. PMID 30241148
- [Background] Shyirambere C, Villaverde C, Nguyen C, Ruhangaza D, Umwizerwa A, Nsanzimana O, Mujyuwisha L, Iradukunda E, Shulman LN, Lehmann L. Nephroblastoma Treatment and Outcomes in a Low-Income Setting. JCO Glob Oncol. 2022 Jul;8:e2200036. doi: 10.1200/GO.22.00036. PMID 35820081
- [Background] Holmes DM, Matatiyo A, Mpasa A, Huibers MHW, Manda G, Tomoka T, Mulenga M, Namazzi R, Mehta P, Zobeck M, Mzikamanda R, Chintagumpala M, Allen C, Nuchtern JG, Borgstein E, Aronson DC, Ozuah N, Nandi B, McAtee CL. Outcomes of Wilms tumor therapy in Lilongwe, Malawi, 2016-2021: Successes and ongoing research priorities. Pediatr Blood Cancer. 2023 May;70(5):e30242. doi: 10.1002/pbc.30242. Epub 2023 Feb 16. PMID 36798020
- [Background] Ravindranath Y, Chang M, Steuber CP, Becton D, Dahl G, Civin C, Camitta B, Carroll A, Raimondi SC, Weinstein HJ; Pediatric Oncology Group. Pediatric Oncology Group (POG) studies of acute myeloid leukemia (AML): a review of four consecutive childhood AML trials conducted between 1981 and 2000. Leukemia. 2005 Dec;19(12):2101-16. doi: 10.1038/sj.leu.2403927. PMID 16136167
- [Background] Hu Y, Chen A, Gao L, He H, Jiang S, Zheng X, Xiao P, Lu J, Wang Y, Li J, Li J, Fan J, Yao Y, Ling J, Fan L, Cheng S, Cheng C, Fang F, Pan J, Wang QF, Ribeiro RC, Hu S. Minimally myelosuppressive regimen for remission induction in pediatric AML: long-term results of an observational study. Blood Adv. 2021 Apr 13;5(7):1837-1847. doi: 10.1182/bloodadvances.2020003453. PMID 33787864
- [Background] Hu Y, Chen A, Zheng X, Lu J, He H, Yang J, Zhang Y, Sui P, Yang J, He F, Wang Y, Xiao P, Liu X, Zhou Y, Pei D, Cheng C, Ribeiro RC, Hu S, Wang QF. Ecological principle meets cancer treatment: treating children with acute myeloid leukemia with low-dose chemotherapy. Natl Sci Rev. 2019 May;6(3):469-479. doi: 10.1093/nsr/nwz006. Epub 2019 Jan 22. PMID 34691895
- [Background] Kapoor A, Beniwal SK, Kalwar A, Singhal MK, Nirban RK, Kumar HS. Metronomic therapy with oral 6-mercaptopurine in elderly acute myeloid leukemia: A prospective pilot study. South Asian J Cancer. 2016 Apr-Jun;5(2):70-2. doi: 10.4103/2278-330X.181644. PMID 27275453
- [Background] Hunger SP, Mullighan CG. Acute Lymphoblastic Leukemia in Children. N Engl J Med. 2015 Oct 15;373(16):1541-52. doi: 10.1056/NEJMra1400972. No abstract available. PMID 26465987
- [Background] Klein K, Haarman EG, de Haas V, Zwaan ChM, Creutzig U, Kaspers GL. Glucocorticoid-Induced Proliferation in Untreated Pediatric Acute Myeloid Leukemic Blasts. Pediatr Blood Cancer. 2016 Aug;63(8):1457-60. doi: 10.1002/pbc.26011. Epub 2016 Apr 19. PMID 27093190
- [Background] McAtee CL, Schneller N, Brackett J, Bernhardt MB, Schafer ES. Treatment-related sinusoidal obstruction syndrome in children with de novo acute lymphoblastic leukemia during intensification. Cancer Chemother Pharmacol. 2017 Dec;80(6):1261-1264. doi: 10.1007/s00280-017-3453-z. Epub 2017 Oct 19. PMID 29051993
- [Background] Bondarenko M, Le Grand M, Shaked Y, Raviv Z, Chapuisat G, Carrere C, Montero MP, Rossi M, Pasquier E, Carre M, Andre N. Metronomic Chemotherapy Modulates Clonal Interactions to Prevent Drug Resistance in Non-Small Cell Lung Cancer. Cancers (Basel). 2021 May 7;13(9):2239. doi: 10.3390/cancers13092239. PMID 34066944
- [Background] Cazzaniga ME, Cordani N, Capici S, Cogliati V, Riva F, Cerrito MG. Metronomic Chemotherapy. Cancers (Basel). 2021 May 6;13(9):2236. doi: 10.3390/cancers13092236. PMID 34066606
- [Background] Minard-Colin V, Auperin A, Pillon M, Burke GAA, Barkauskas DA, Wheatley K, Delgado RF, Alexander S, Uyttebroeck A, Bollard CM, Zsiros J, Csoka M, Kazanowska B, Chiang AK, Miles RR, Wotherspoon A, Adamson PC, Vassal G, Patte C, Gross TG; European Intergroup for Childhood Non-Hodgkin Lymphoma; Children's Oncology Group. Rituximab for High-Risk, Mature B-Cell Non-Hodgkin's Lymphoma in Children. N Engl J Med. 2020 Jun 4;382(23):2207-2219. doi: 10.1056/NEJMoa1915315. PMID 32492302
- [Background] van Weelderen RE, Wijnen NE, Njuguna F, Klein K, Vik TA, Olbara G, Kaspers GJL. Treatment outcomes of pediatric acute myeloid leukemia in Western Kenya before and after the implementation of the SIOP PODC treatment guideline. Cancer Rep (Hoboken). 2023 Aug;6(8):e1849. doi: 10.1002/cnr2.1849. Epub 2023 Jun 22. PMID 37349659
- [Background] Gallegos-Castorena S, Medina-Sanson A, Gonzalez-Ramella O, Sanchez-Zubieta F, Martinez-Avalos A. Improved treatment results in Mexican children with acute myeloid leukemia using a Medical Research Council (MRC)-acute myeloid leukemia 10 modified protocol. Leuk Lymphoma. 2009 Jul;50(7):1132-7. doi: 10.1080/10428190902964768. PMID 19557634
- [Background] Howard SC, Davidson A, Luna-Fineman S, Israels T, Chantada G, Lam CG, Hunger SP, Bailey S, Ribeiro RC, Arora RS, Pedrosa F, Harif M, Metzger ML. A framework to develop adapted treatment regimens to manage pediatric cancer in low- and middle-income countries: The Pediatric Oncology in Developing Countries (PODC) Committee of the International Pediatric Oncology Society (SIOP). Pediatr Blood Cancer. 2017 Dec;64 Suppl 5. doi: 10.1002/pbc.26879. PMID 29297619
- [Background] Parikh NS, Howard SC, Chantada G, Israels T, Khattab M, Alcasabas P, Lam CG, Faulkner L, Park JR, London WB, Matthay KK; International Society of Pediatric Oncology. SIOP-PODC adapted risk stratification and treatment guidelines: Recommendations for neuroblastoma in low- and middle-income settings. Pediatr Blood Cancer. 2015 Aug;62(8):1305-16. doi: 10.1002/pbc.25501. Epub 2015 Mar 21. PMID 25810263
- [Background] Bouda GC, Traore F, Couitchere L, Raquin MA, Guedenon KM, Pondy A, Moreira C, Rakotomahefa M, Harif M, Patte C. Advanced Burkitt Lymphoma in Sub-Saharan Africa Pediatric Units: Results of the Third Prospective Multicenter Study of the Groupe Franco-Africain d'Oncologie Pediatrique. J Glob Oncol. 2019 Nov;5:1-9. doi: 10.1200/JGO.19.00172. PMID 31794283
- [Background] Bansal D, Davidson A, Supriyadi E, Njuguna F, Ribeiro RC, Kaspers GJL. SIOP PODC adapted risk stratification and treatment guidelines: Recommendations for acute myeloid leukemia in resource-limited settings. Pediatr Blood Cancer. 2023 Nov;70(11):e28087. doi: 10.1002/pbc.28087. Epub 2019 Nov 27. PMID 31774234
- [Background] Israels T, Moreira C, Scanlan T, Molyneux L, Kampondeni S, Hesseling P, Heij H, Borgstein E, Vujanic G, Pritchard-Jones K, Hadley L. SIOP PODC: clinical guidelines for the management of children with Wilms tumour in a low income setting. Pediatr Blood Cancer. 2013 Jan;60(1):5-11. doi: 10.1002/pbc.24321. Epub 2012 Sep 26. PMID 23015404
- [Background] Espinoza D, Blanco Lopez JG, Vasquez R, Fu L, Martinez R, Rodriguez H, Navarrete M, Howard SC, Friedrich P, Valsecchi MG, Conter V, Ceppi F. How should childhood acute lymphoblastic leukemia relapses in low-income and middle-income countries be managed: The AHOPCA-ALL study group experience. Cancer. 2023 Mar 1;129(5):771-779. doi: 10.1002/cncr.34572. Epub 2022 Dec 12. PMID 36504077
- [Background] van Weelderen RE, Njuguna F, Klein K, Mostert S, Langat S, Vik TA, Olbara G, Kipng'etich M, Kaspers GJL. Outcomes of pediatric acute myeloid leukemia treatment in Western Kenya. Cancer Rep (Hoboken). 2022 Oct;5(10):e1576. doi: 10.1002/cnr2.1576. Epub 2021 Nov 22. PMID 34811958
- [Background] Kersten E, Scanlan P, Dubois SG, Matthay KK. Current treatment and outcome for childhood acute leukemia in Tanzania. Pediatr Blood Cancer. 2013 Dec;60(12):2047-53. doi: 10.1002/pbc.24576. Epub 2013 Aug 26. PMID 24039163
- [Background] Ngwa W, Addai BW, Adewole I, Ainsworth V, Alaro J, Alatise OI, Ali Z, Anderson BO, Anorlu R, Avery S, Barango P, Bih N, Booth CM, Brawley OW, Dangou JM, Denny L, Dent J, Elmore SNC, Elzawawy A, Gashumba D, Geel J, Graef K, Gupta S, Gueye SM, Hammad N, Hessissen L, Ilbawi AM, Kambugu J, Kozlakidis Z, Manga S, Maree L, Mohammed SI, Msadabwe S, Mutebi M, Nakaganda A, Ndlovu N, Ndoh K, Ndumbalo J, Ngoma M, Ngoma T, Ntizimira C, Rebbeck TR, Renner L, Romanoff A, Rubagumya F, Sayed S, Sud S, Simonds H, Sullivan R, Swanson W, Vanderpuye V, Wiafe B, Kerr D. Cancer in sub-Saharan Africa: a Lancet Oncology Commission. Lancet Oncol. 2022 Jun;23(6):e251-e312. doi: 10.1016/S1470-2045(21)00720-8. Epub 2022 May 9. PMID 35550267
- [Background] Creutzig U, Zimmermann M, Bourquin JP, Dworzak MN, Fleischhack G, Graf N, Klingebiel T, Kremens B, Lehrnbecher T, von Neuhoff C, Ritter J, Sander A, Schrauder A, von Stackelberg A, Stary J, Reinhardt D. Randomized trial comparing liposomal daunorubicin with idarubicin as induction for pediatric acute myeloid leukemia: results from Study AML-BFM 2004. Blood. 2013 Jul 4;122(1):37-43. doi: 10.1182/blood-2013-02-484097. Epub 2013 May 23. PMID 23704089
- [Background] Begum M, Islam A, Rahman AA, Akter M, Alam ST, Tasmeen R. Abandonment and Outcome of Childhood Acute Myeloid Leukemia in A Tertiary Level Hospital. Mymensingh Med J. 2018 Jan;27(1):95-102. PMID 29459598
- [Background] N, H. et al. SEER Cancer Statistics Review, 1975-2017. SEER Cancer Statistics Review, 1975-2017, National Cancer Institute.